CLINICAL TRIAL: NCT05764876
Title: Repurposing Clinically Approved Drugs for Yaws with an Insight Into the Cutaneous Ulcer Disease Syndrome (Trep-AByaws)
Acronym: Trep-AByaws
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fundación FLS de Lucha Contra el Sida, las Enfermedades Infecciosas y la Promoción de la Salud y la Ciencia (Other)
Collaborators: National Department of Health, Papua New Guinea (Unknown); School of Medicine and Health Sciences, University of Papua New Guinea (Unknown)
Responsible Party: Principal Investigator, Oriol Mitja, Associate Professor, Infectious Diseases and Global Health, Fundación FLS de Lucha Contra el Sida, las Enfermedades Infecciosas y la Promoción de la Salud y la Ciencia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Trep-AByaws
Record Dates: First submitted 2023-02-02; First posted 2023-03-13 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2024-07

CONDITIONS: Yaws; Cutaneous Ulcer
Keywords: azithromycin; linezolid
MeSH Terms: conditions — Yaws; Skin Ulcer | interventions — Linezolid; Azithromycin

STUDY DESIGN:
Intervention Model Description: Open-label, non inferiority, two arms and randomized clinical trial. Eligible patients will be randomized (1:1) to receive Linezolid (experimental arm) or Azithromycin (control arm).
Who Masked: Investigator
Masking Description: Investigator will not be present for treatment nor for outcome assessment, and data analysis (statistics) will be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Azithromycin (Active Comparator): Participants in the control arm will receive standard treatment for yaws which azithromycin .
  Interventions: Drug: Azithromycin Oral Tablet
- Linezolid (Experimental): Participants in the experimental arm will receive oral linezolid treatment.
  Interventions: Drug: Linezolid Oral Tablet

INTERVENTIONS:
Drug: Linezolid Oral Tablet — Oral tablet of linezolid 10mg/kg every 8 hours for 7 days.
  Other Names: Zyvox, Zyvoxid
  Arms: Linezolid
Drug: Azithromycin Oral Tablet — Oral tablet of azithromycin 30mg/kg maximum 2gr single dose.
  Other Names: Zithromax
  Arms: Azithromycin

SUMMARY:
The goal of this clinical trial is to test the non inferiority of linezolid compared with azithromycin as a treatment for yaws . The main questions it aims to answer are: can linezolid cure active yaws, and can linezolid cure latent yaws. Participants with serologically confirmed yaws will be randomized to receive linezolid (experimental) or azithromycin (control group) treatment and followed up to assess clinical resolution.

DETAILED DESCRIPTION:
The current principle of yaws eradication is based on a single round of mass drug administration of azithromycin (AZI) called total community treatment (TCT) followed by targeted treatment of active cases and close contacts every 6 months called total targeted treatment (TTT). Studies done in Papua New Guinea have shown that 3 rounds of TCT are preferable to 1 TCT followed by TTT rounds because it results in higher overall coverage, particularly of latent cases. In the context of repeated rounds of TTT and multiple rounds of TCT, resistance to AZI has ben detected on 5 patients with yaws Recent studies have been successful on the culture of Treponema pallidum (syphilis and yaws), therefore investigators are now able to identify more potential treatment for yaws and syphilis.

Yaws is one of the major causes of the Cutaneous Ulcer Disease (CUD) syndrome. The CUD syndrome is a painful and debilitating condition, endemic to remote tropical regions with poor sanitation and limited health care access affecting children mainly. In Papua New Guinea it is caused by a range of unknown and some known pathogens besides yaws that are not easily distinguished on clinical diagnosis. New information on the causative agents of the CUD syndrome is needed to facilitate its management with an integrated approach.

The aim of the project is to provide evidence supporting (or rejecting) the hypothesis that the use of linezolid (LZD) can be an alternative treatment to cure yaws corroborated by clinical, serological, and molecular methods. LZD is a very safe drug that has been delivered to adults and children for the treatment of cutaneous infections all over the world. Investigators will compare two different treatments: (A) linezolid (LZD) and (B) azithromycin (AZI). In addition, the investigators plan to contribute to characterize the etiology of the CUD syndrome. The study will be implemented in selected wards of the Islands Region of Papua New Guinea.

ELIGIBILITY:
Inclusion Criteria:

1. Participants 5-18 years identified during an active case search program at the elementary, primary and secondary schools in the Islands Region.
2. CUD syndrome suspected due to yaws: one or more ulcerative or nodular or papilloma skin lesion of more than 1 cm in diameter.
3. Positive treponemal (T1) and non-treponemal (T2) serology by Chembio dual path platform (DPP) syphilis screen & confirm assay (DPP test).
4. Accepted and signed informed consent.
5. Ability to comply with the requirements of the study protocol including follow up visits.

Exclusion Criteria:

1. Children younger than 5 years old.
2. Clinical late-stage possible yaws: destructive osteitis (rhinopharyngitis gangosa, sabre shins) or gummous nodules.
3. Known allergy to LZD or AZI antibiotics.
4. Pregnant or breastfeeding women.
5. Refusal at ward level or village chief (for village inclusion), or refusal of individual or guardian (for individual inclusion).
6. Have taken any antibiotics with potential activity against TPE within the last 7 days prior to randomization (i.e., beta lactams, cephalosporines, macrolides, tetracyclines).
7. Uncontrolled hypertension, pheochromocytoma, thyrotoxicosis, carcinoid syndrome, bipolar disorder, incapacitating psycho-affective disturbance, acute confusional state.
8. Renal function impairment requiring hemodialysis.
9. Current treatment with any drugs likely to interact with the study medication
10. Symptomatic concomitant infection requiring antibiotic treatment potentially active against TPE.
11. Having received treatment for yaws in the last 6 months.
12. Patients who are unable to take oral medication or having a gastrointestinal disease likely to interfere with drug absorption (including malnutrition and stomach flu).

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 465 (Actual)
Dates: Start 2023-03-14 (Actual); Primary Completion 2024-06-20 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Clinical resolution | 4 weeks after treatment
  Proportion of patients with clinical resolution of yaws lesions (clinical cure). Assessment of clinical resolution defined as the complete healing of lesions at 4 weeks from treatment start.
Serological cure | 24 weeks after treatment
  Proportion of patients with adequate serological response (serological cure). Assessment of sero-cure is described as a four-fold decline in rapid plasma reagin (RPR) titer or seroreversion at 24 weeks from treatment start.
Serological cure | 48 weeks after treatment
  Proportion of patients with adequate serological response (serological cure). Assessment of sero-cure is described as a four-fold decline in rapid plasma reagin (RPR) titer or seroreversion at 48 weeks from treatment start.
Relapse | 24 weeks after treatment
  Proportion of patients with relapse (recurrent episodes caused by the same strain) (molecular cure). Assessment of recurrence by molecular methods of Treponema pallidum ssp. pertenue (TPE) DNA in ulcer swab to determine relapse or reinfection within 24 weeks from treatment start.
Relapse | 48 weeks after treatment
  Proportion of patients with relapse (recurrent episodes caused by the same strain) (molecular cure). Assessment of recurrence by molecular methods of Treponema pallidum ssp. pertenue (TPE) DNA in ulcer swab to determine relapse or reinfection within 48 weeks from treatment start.

SECONDARY OUTCOMES:
Lession (ulcer swab) TPE assessment | Baseline (before treatment)
  Assessment of TPE strains by genomic molecular methods in ulcer swabs from patients with active yaws.
Oral (oral swab) TPE assessment | Baseline (before treatment)
  Assessment of TPE strains by genomic molecular methods in oral swabs from patients with active/latent yaws.
Plasma TPE assessment | Baseline (before treatment)
  Assessment of TPE strains by genomic molecular methods in plasma from patients with active/latent yaws.
Allelic variation in recurrent cases | Baseline (before treatment)
  Proportion of patients with allelic variation in TPE DNA in patients with recurrence or treatment failure.
Identification of antibiotic resistance genotype. | 4 weeks after treatment
  Proportion of patients with antibiotic resistance genotype.
Identification of other causes of cutaneous ulcer | Baseline (before treatment)
  Proportion of patients with selected known and unknown causes of cutaneous ulcers (CU). Assessment of etiological agents using polymerase chain reaction (PCR) for TPE, Haemophylus ducreyi (HD) and Streptoccocus pyogenes (SP).
Safety of intervention (adverse events) | 48 weeks after treatment.
  Proportion of patients with adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Camila Beiras, Study Director — Fundació Lluita contra les Infeccions
Locations (1):
- National Department of Health, Port Moresby, Papua New Guinea

IPD SHARING:
Plan to Share IPD: Undecided
Protocol and anonymised data will be made available upon reasonable request